CLINICAL TRIAL: NCT05358743
Title: Effect of Probiotics on Oral Candida Colonization Level in Complete Denture Wearers (Randomized Controlled Clinical Trial)
Brief Title: Effect of Probiotics on Oral Candida Among Denture Wearers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: probiotics_2022
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Oral Candida Albicans Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental)
  Interventions: Other: Probiotic group
- Control group (Placebo Comparator)
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: Probiotic group — Participants will use the probiotic product once daily (1 tablet/day) for 8 weeks
  Arms: Probiotic group
Other: Placebo group — Patients will chew placebo products (blueberry tablets) once daily (1 tablet/day) for 8 weeks.
  Arms: Control group

SUMMARY:
Forty-eight denture wearers with detectable levels of candida colonization without clinical symptoms will be randomly allocated into two groups: probiotics and placebo. All patients will take a daily dose of chewable tablets (probiotics or placebo according to the assigned group) for 8 weeks. Samples of mouth rinse will be collected from patients at baseline, 4 weeks from the beginning of the intervention, 8 weeks (the end of intervention), and after another 4 weeks for post-intervention follow up. Samples will be tested for both candida count and candida species identification

ELIGIBILITY:
Inclusion Criteria:

* Detectable levels of Candida in palatal mucosa without clinical symptoms of active candidiasis.
* Completely edentulous arches with newly formed denture .
* Patients with controlled hypertension, and diabetes will be included in this study as they are considered very common problems in the targeted population.

Exclusion Criteria:

* Inability to understand/ follow the experimental procedures,
* Administration of topic or systemic antifungal or antibacterial agents in the previous 60 days.
* Consumption of probiotics.
* GITdisorders.
* Heartdisease.
* Diseases that significantly influence immunity such as; kidney problems, head and neck cancer, or radiotherapy, AIDS, or immunosuppressive therapy.
* Clinical manifestations of oral candidiasis.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in candida count | Baseline, 4 weeks, 8 weeks, 12 weeks
  Quantitative culture will be performed from mouth-rinse samples by inoculation onto the surface of Sabouraud dextrose agar plates with chloramphenicol, and subsequent aerobic incubation for 24 to 48 hours at 37°C.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt